CLINICAL TRIAL: NCT01175707
Title: A Phase 4, Prospective, Randomized, Open-label Study to Compare Use of Cubicin With Vancomycin Administered Intravenously in the Treatment of Patients With Complicated Skin and Skin Structure Infections Due to Suspected or Confirmed Gram-positive Bacteria in a Home Infusion Setting
Brief Title: Study Comparing Cubicin With Vancomycin in Treatment of Participants With Complicated Skin and Skin Structure Infections in a Home Infusion Setting
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Business decision
Sponsor: Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 3009-009; DAP-4HOME-09-05 (Other: Cubist Study Number)
Record Dates: First submitted 2010-07-20; First posted 2010-08-05 (Estimated); Results first posted 2015-05-13 (Estimated); Last update posted 2018-12-26 (Actual); Status verified 2018-12

CONDITIONS: Complicated Skin or Skin Structure Infection
MeSH Terms: interventions — Daptomycin; Vancomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Daptomycin (Experimental): 500 milligrams (mg) daptomycin, administered intravenously (IV) for 7 to 10 days accordingly to the package insert or according to institutional practice, if warranted
  Interventions: Drug: Daptomycin
- Vancomycin (Active Comparator): Vancomycin monotherapy is administered according to prescribing physician's order with duration of treatment modified, if warranted, according to Investigator site's standard practice, and End of Treatment (EOT) is dependent on this. Dose adjustments of vancomycin will be suggested by the pharmacist and approved by prescribing or following physician
  Interventions: Drug: Vancomycin

INTERVENTIONS:
Drug: Daptomycin
  Other Names: Cubicin
  Arms: Daptomycin
Drug: Vancomycin
  Arms: Vancomycin

SUMMARY:
This is a randomized, open-label, multi-center, phase 4 study designed to compare intravenous (IV) daptomycin and IV vancomycin administered in a home infusion setting for the treatment of complicated skin and skin structure infections (cSSSI) due to Gram-positive bacteria in participants who are prescribed vancomycin for 7 to 14 days and who are planning to receive vancomycin in a home-infusion setting.

DETAILED DESCRIPTION:
This is a randomized, open-label, multi-center, phase 4 study. The overall goals of this study are to compare intravenous (IV) daptomycin and IV vancomycin administered in a home infusion setting for the treatment of cSSSI due to Gram-positive bacteria in participants who are prescribed vancomycin for 7-14 days and who are planning to receive vancomycin in a home infusion setting. Study objectives include evaluation of clinical and resource utilization endpoints and economic analysis from the perspective of the home infusion provider.

ELIGIBILITY:
Inclusion Criteria:

* Complicated skin or skin structure infection (cSSSI)
* Intravenous vancomycin home infusion ordered for 7-14 days

Exclusion Criteria:

* Pregnant or lactating female
* Concurrently receiving other systemic antibiotics with gram positive activity
* Known or suspected allergy or hypersensitivity to daptomycin or vancomycin
* Known or suspected vancomycin-resistant enterococci (VRE)
* Known or suspected osteomyelitis, pneumonia, bacteremia, endocarditis, or urinary tract infection
* Known or suspected human immunodeficiency virus (HIV), cancer, or autoimmune disease such as lupus
* Receiving systemic concomitant immunosuppressive agents such as chemotherapy, corticosteroids, tacrolimus, sirolimus, or cyclosporine, during the duration of the study
* Requirement for non-study gram positive systemic antibiotics
* Known to be allergic or intolerant to intravenous vancomycin or daptomycin
* Participants with known or suspected creatinine clearance (CLcr) < 30 milliliters per minute (mL/min)
* In skilled nursing facility
* In hospice or admission to hospice is planned

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2010-07-15 (Actual); Primary Completion 2011-11-17 (Actual); Study Completion 2011-11-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paula Bokesch, MD, Study Director — Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA)
Locations (4):
- United States (4):
  - Heartland I.V. Care, Livonia, Michigan
  - Heartland I.V. Care, Roseville, Minnesota
  - Heartland I.V. Care, Pittsburgh, Pennsylvania
  - NationsMed Clinical Research, Inc., Stafford, Texas

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Daptomycin | Vancomycin
Started | 40 | 40
Completed | 36 | 34
Not Completed | 4 | 6
Not completed — Adverse Event | 4 | 6

BASELINE CHARACTERISTICS:
Population: All study participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Daptomycin | Vancomycin | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.55 (14.387) | 56.78 (19.366) | 57.665 (16.8765)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 21 | 40
  Male | 21 | 19 | 40

OUTCOME MEASURES:

1. Primary Outcome: Time Spent (Minutes) for Home Infusion Therapy
Description: Each participant is counted once per category. Avg=average; Admin=administer.
Time Frame: Day 1 up to Day 14
Population: All study participants.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Daptomycin | Vancomycin
Number analyzed (Participants) | 40 | 40
Minutes
  Total antibiotic therapy duration | 160.7 (326.07) | 1430.1 (1331.45)
  Total time to administer drug | 87.6 (132.66) | 1001.7 (696.76)
  Avg time per day to administer drug | 6.64 (8.221) | 127.78 (59.565)
  Avg time to admin drug per infusion | 6.64 (8.221) | 95.81 (23.566)
  Total caregiver time to admin drug | 261.8 (494.86) | 1336 (1527.67)
  Avg caregiver time per day to admin drug | 16.66 (21.376) | 148.66 (174.709)
  Avg caregiver time per infusion to admin drug | 16.66 (21.376) | 124.25 (175.856)
  Total nursing time | 393.0 (229.34) | 404.2 (321.42)
  Avg nursing time per visit | 73.25 (17.920) | 85.80 (23.907)
  Avg nursing time per day | 73.97 (17.759) | 87.79 (25.382)
  Total time for pharmacist consultations | 60.4 (29.59) | 55.3 (35.67)

2. Primary Outcome: Total Antibiotic Therapy Duration (in Days) Per Participant for Home Infusion Therapy
Description: The mean duration in home-infusion antibiotic therapy per participant is presented.
Time Frame: Day 1 up to Day 14
Population: All study participants.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Daptomycin | Vancomycin
Number analyzed (Participants) | 40 | 40
Days | 13.0 (6.05) | 11.0 (6.11)

3. Primary Outcome: Number of Nurse Visits or Consultations Per Participant for Home Infusion Therapy
Description: Each participant is counted once per category.
Time Frame: Day 1 up to Day 14
Population: All study participants.
Measure: Mean (Standard Deviation); unit: Visits or Consultations per Participant
Arm/Group | Daptomycin | Vancomycin
Number analyzed (Participants) | 40 | 40
Visits or Consultations per Participant
  Total number of nursing visits | 5.8 (3.90) | 5.0 (4.18)
  Total number of scheduled nursing visits | 4.1 (1.91) | 4.4 (3.98)
  Total number of unscheduled nursing visits | 4.91 (4.0) | 1.24 (1.0)
  Total number of pharmacist consultations | 9.6 (4.22) | 9.6 (5.79)

4. Primary Outcome: Number of Participants With at Least 1 Unscheduled Nursing Visit During Home Infusion Therapy
Time Frame: Day 1 up to Day 14
Population: Number of Participants Analyzed based on number of participants with at least one nurse visit/pharmacist consultation within each treatment group results in 39 participants analyzed for the Daptomycin ARM group for this Outcome Measure.
Measure: Number; unit: Participants
Arm/Group | Daptomycin | Vancomycin
Number analyzed (Participants) | 39 | 40
Participants | 12 | 15

5. Primary Outcome: Number of Participants With at Least One Pharmacist Consultation During Home Infusion Therapy
Time Frame: Day 1 up to Day 14
Population: All study participants.
Measure: Number; unit: Participants
Arm/Group | Daptomycin | Vancomycin
Number analyzed (Participants) | 40 | 40
Participants | 40 | 40

6. Primary Outcome: Reasons for Nurse Visits During Home Infusion Therapy
Description: The reason for a participant's nurse visit is presented. There may be more than one reason for nurse visits per participant.
Time Frame: Day 1 up to Day 14
Population: All study participants.
Measure: Number; unit: Reason Cited
Arm/Group | Daptomycin | Vancomycin
Number analyzed (Participants) | 40 | 40
Reason Cited
  Laboratory assessment | 36 | 36
  Participant/Caregiver teaching | 26 | 29
  Site/Catheter care | 5 | 10
  Clinical assessment | 1 | 2
  Other | 28 | 19

7. Primary Outcome: Reasons for Pharmacist Consultations During Home Infusion Therapy
Description: The reason for a participant's pharmacist consultation is presented. There may be more than one reason for pharmacist consultations per participant.
Time Frame: Day 1 up to Day 14
Population: All study participants.
Measure: Number; unit: Reason Cited
Arm/Group | Daptomycin | Vancomycin
Number analyzed (Participants) | 40 | 40
Reason Cited
  Development/revision of care plan | 25 | 25
  Review of written reports of participant status | 16 | 20
  Review of related labs and other studies | 38 | 36
  Communication - participant | 38 | 37
  Communication - prescriber | 26 | 25
  Communication - home care nurse | 25 | 20
  Communication - integration of new information | 3 | 4
  Other | 13 | 13

8. Primary Outcome: Percentage of Treatment Goals Met at End of Therapy
Description: Treatment goals included: 1. Elimination of infection/achieved desired response. 2. Laboratory values were within normal limits or improved indicating progress toward therapy goal. 3. Pain was controlled. 4. Participant did not have catheter site complications (eg,infection, loss of patency). 5. Participant had no knowledge deficits related to administration, equipment use, side effects and waste disposal. 6. Participant had no side effects, adverse drug reactions and/or drug or food interactions. 7. Signs and symptoms of infection did improve or resolve. 8. Participant was compliant with IV therapy 9. Successfully completed therapy without interruptions, unexpected hospitalizations. 10. Participant continued on an oral antibiotic. 11. Participant continued on an IV antibiotic.
  Each participant's percentage was derived from number of treatment goals achieved out of a maximum of 11 goals. Reported percentage below is the average of all participants' percentage of goals met by arm.
Time Frame: Day 1 up to Day 14
Population: All study participants.
Measure: Mean (Standard Deviation); unit: Percentage of Goals Met
Arm/Group | Daptomycin | Vancomycin
Number analyzed (Participants) | 40 | 40
Percentage of Goals Met | 74.98 (10.842) | 75.21 (11.823)

9. Secondary Outcome: Number of Participants With at Least 1 Intervention Related to Complicated Skin or Skin Structure Infection (cSSSI) During Home Infusion Therapy
Description: Type of interventions include Intravenous (IV) line replacement, IV line removal, IV line placement (post study therapy), Incision and drainage (wound), Incision and drainage (line), Debridement, Declotting procedure, and Blood draw.
Time Frame: Day 1 up to Day 14
Population: All study participants.
Measure: Number; unit: Participants
Arm/Group | Daptomycin | Vancomycin
Number analyzed (Participants) | 40 | 40
Participants
  Had at least 1 intervention | 9 | 4
  Had no intervention | 31 | 36

10. Secondary Outcome: Mean Number of Interventions Per Participant During Home Infusion Therapy
Description: Type of interventions include IV line replacement, IV line removal, IV line placement (post study therapy), incision and drainage (wound), incision and drainage (line), debridement, declotting procedure, and blood draw.
Time Frame: Day 1 up to Day 14
Population: All study participants.
Measure: Mean (Standard Deviation); unit: Interventions
Arm/Group | Daptomycin | Vancomycin
Number analyzed (Participants) | 40 | 40
Interventions | 1.8 (1.30) | 1.5 (0.58)

11. Secondary Outcome: Number of Intervention Types During Home Infusion Therapy
Description: There may be more than one type of intervention per participant. A participant is counted only once for each category even if they had several instances of a given intervention.
Time Frame: Day 1 up to Day 14
Population: All study participants
Measure: Number; unit: participants
Arm/Group | Daptomycin | Vancomycin
Number analyzed (Participants) | 40 | 40
participants
  IV line replacement | 2 | 0
  Incision and drainage (wound) | 0 | 1
  De-clotting procedure | 3 | 2
  Other | 6 | 2

12. Secondary Outcome: Participants Who Had More Than 1 Laboratory Assessment During Home Infusion Therapy
Description: Laboratory assessments include serum creatinine, creatine phosphokinase (CPK), and Vancomycin trough.
Time Frame: Day 1 up to Day 14
Population: All study participants.
Measure: Number; unit: Participants
Arm/Group | Daptomycin | Vancomycin
Number analyzed (Participants) | 40 | 40
Participants | 40 | 40

13. Secondary Outcome: Mean Number of Laboratory Assessments Per Participant During Home Infusion Therapy
Description: Laboratory assessments include serum creatinine, creatine phosphokinase (CPK), and vancomycin trough.
Time Frame: Day 1 up to Day 14
Population: All study participants.
Measure: Mean (Standard Deviation); unit: Assessments
Arm/Group | Daptomycin | Vancomycin
Number analyzed (Participants) | 40 | 40
Assessments | 2.7 (1.19) | 2.8 (1.24)

14. Secondary Outcome: Number of Laboratory Assessment Types During Home Infusion Therapy
Description: There may be more than one type of laboratory assessment per participant. A participant is counted only once for each category. Laboratory assessments include serum creatinine, creatine phosphokinase (CPK), and vancomycin trough
Time Frame: Day 1 up to Day 14
Population: All study participants.
Measure: Number; unit: Assessments
Arm/Group | Daptomycin | Vancomycin
Number analyzed (Participants) | 40 | 40
Assessments
  Serum creatinine | 40 | 40
  CPK | 39 | 0
  Vancomycin | 1 | 38

15. Secondary Outcome: Health Economic Outcomes in United States (US) Dollars for Home Infusion Therapy Per Participant
Description: Total Heartland costs per participant were derived by summing the costs of drug, pharmacy services/supplies and nursing.
Time Frame: Day 1 up to Day 14
Population: All study participants.
Measure: Mean (Standard Deviation); unit: US Dollars
Arm/Group | Daptomycin | Vancomycin
Number analyzed (Participants) | 40 | 40
US Dollars
  Total Drug Costs | 2762.37 (1446.140) | 107.14 (69.264)
  Pharmacy Service and Supplies Costs | 641.25 (247.263) | 596.25 (278.472)
  Nursing Costs | 637.63 (404.868) | 583.02 (475.495)
  Total Heartland Costs | 3956.25 (1781.020) | 1273.02 (667.673)
  Emergency Room (ER) Visit Costs | 1660.31 (761.630) | 1518 (533.370)
  Lost Work Costs | 3729.13 (3753.586) | 3635.60 (6404.213)

ADVERSE EVENTS:
Arm/Group | Daptomycin | Vancomycin
Serious Adverse Events (participants affected / at risk) | 7/40 | 7/40
Other Adverse Events (participants affected / at risk) | 13/40 | 5/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Daptomycin (N=40) | Vancomycin (N=40)
Infection (Infections and infestations) | 2 | 3
Cellulitis (Infections and infestations) | 2 | 1
Device related infection (Infections and infestations) | 0 | 1
Gangrene (Infections and infestations) | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Blood creatinine increased (Investigations) | 0 | 1
White blood cell count increased (Investigations) | 0 | 1
Gout (Metabolism and nutrition disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Daptomycin (N=40) | Vancomycin (N=40)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 1 (1)
Catheter site erythema (General disorders) | 1 (1) | 0 (0)
Catheter site haemorrhage (General disorders) | 1 (2) | 0 (0)
Device occlusion (General disorders) | 1 (1) | 0 (0)
Infusion site pain (General disorders) | 1 (1) | 0 (0)
Medical device complication (General disorders) | 2 (2) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Abscess (Infections and infestations) | 1 (1) | 0 (0)
Breast cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 2 (3) | 0 (0)
Fungal infection (Infections and infestations) | 1 (1) | 0 (0)
Fungal skin infection (Infections and infestations) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was terminated prematurely.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first publication is initiated by Cubist. If First Publication not published within 1 year of Study conclusion or termination, Investigator has right to publish and disclose the Data. Prior to any submission for publication, presentation, or communication of results or information arising from the Study, Investigator shall provide Cubist at least 90 days for review and comment upon the manuscript or other material for such publication or presentation.